CLINICAL TRIAL: NCT03352752
Title: The Effect of Virtual Reality Technology to Alleviate the Acute Pain of Scar Treatment With Fractional Laser Under Local Anesthesia: a Single Center, Randomized, Controlled, Clinical Study
Brief Title: Virtual Reality Technology to Alleviate the Acute Pain of Scar Treatment With Fractional Laser Under Local Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kai-Yang Lv (Other)
Responsible Party: Sponsor-Investigator, Kai-Yang Lv, Associate Professor, Changhai Hospital
Organization: Changhai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: kylv
Record Dates: First submitted 2017-11-17; First posted 2017-11-24 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Scar; Acute Pain
Keywords: virtual reality; fractional laser; scars; acute pain; anxiety score
MeSH Terms: conditions — Cicatrix; Acute Pain

STUDY DESIGN:
Intervention Model Description: It's a randomized controlled study, there were 218 cases, the ratio of the control group to the experimental group was one to one，109 cases per group.
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Possess HTC Vive before the operation (Experimental): The experimental group was wearing VR helmet before operation, and the immersion experience was selected from the video content library pre-selected. After 3 minutes of the VR experience, the surgeon started the fractional laser operation (Notify the patient). The operating area is continuous 10 maximum square spot areas.The parameters for the DEEP FX mode:35mj, 5% density, 300Hz.
  Interventions: Device: HTC Vive
- Without HTC Vive before the operation (Experimental): The control group was wearing a blindfold before operation. The operating area is continuous 10 maximum square spot areas. The parameters for the DEEP FX mode:35mj, 5% density, 300Hz.
  Interventions: Other: Without HTC Vive

INTERVENTIONS:
Device: HTC Vive — Wearing VR helmet before operation
  Arms: Possess HTC Vive before the operation
Other: Without HTC Vive — Wearing a blindfold before operation
  Arms: Without HTC Vive before the operation

SUMMARY:
This study evaluates the effect of virtual reality technology alleviates the acute pain of scar treatment with fractional laser under local anesthesia

DETAILED DESCRIPTION:
Fractional laser surgery under local anesthesia will accompany by the pain and anxiety. It's a bad experience for the patients. The effect of Virtual Reality (virtual reality, VR) to alleviate pain and anxiety of fractional laser treatment of scar is still not studied. Virtual reality technology is an important direction of simulation technology. Including the computer graphics technology, human-computer interface technology, multimedia technology, sensor technology, network technology and other collection technology. Usually generated by a real-time 3D animation of the computer system, a location tracker data. The handle and the head mounted display technology is commonly used in a variety of clinical invasive procedures, such as debridement and burn patients physical therapy, dental pain, injection pain, chronic itching. Previous study shows that VR as a distraction therapy, compared to the traditional methods ,for example watching video and listening to music, has stronger individual initiative and human-computer interaction, it shows a stronger analgesic effect.

HTC Vive is a VR headset, jointly developed by HTC company and Valve company. This equipment could improve the virtual reality experience and bring obvious analgesic effect. There are reasons to believe that HTC Vive could bring the best immersion experience and could be obviously decrease pain and anxiety of scar treatment with fractional laser under local anesthesia.

This study was conducted at department of burn, Changhai hospital, and all operations completed by experienced surgeons (researcher).

This study is a prospective randomized controlled study. A group of patients wear a blindfold and the other group treated with VR equipment (HTC Vive) after localized anesthesia with standard lidocaine cream. Finally, the differences of pain score,anxiety score, physiological indicators and satisfaction between two groups are compared. This study could provide a safe and non-drug intervention measure for patients receive fractional laser treatment under local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant women between the ages of 18 and 60；
2. The scar site to be treated is located outside the head and face, scar area ≥ 0.5% total body surface area (TBSA)；
3. All patients should be sign information.

Exclusion Criteria:

1. Poor physical condition before operative, it is estimated that can't tolerate local anesthesia surgery；
2. Associated with malignant tumors, all kinds of heart disease history, hypertensive patients;
3. Patients with mental illness, alcohol-dependent patients, post-traumatic stress disorder, drug abuse history, and drug addicts; patients with pregnancy; lidocaine cream allergies;
4. Patients can't tolerate VR experience or participate in other clinical trials；
5. Unable or unwilling to comply with research programs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 218 (Estimated)
Dates: Start 2017-08-02 (Actual); Primary Completion 2020-08-11 (Estimated); Study Completion 2020-12-21 (Estimated)

PRIMARY OUTCOMES:
Pain scores | From before the operation to the end the surgery; about one hour
  Intraoperative pain score, postoperation pain score.(0: no pain; 10: worst imaginable pain)

SECONDARY OUTCOMES:
Anxiety score | From beginning of the operation to the end of the operation; about one hour
  Intraoperative anxiety score, preoperative anxiety score.
Heart rate | From into the group to the end of the surgery;about six hours
  Intraoperative highest heart rate, preoperative heart rate and postoperative heart rate.
Respiratory rate | From into the group to the end of the surgery;about six hours
  Preoperative respiratory rate, intraoperative maximum respiratory rate and postoperative respiratory rate.
Blood pressure | From the into the group to the end of the surgery;about six hours
  Preoperative basal blood pressure and postoperative blood pressure.
Surgical satisfaction | From beginning of the operation to the end of the operation;about one hour
  Surgical satisfaction of treatment with 10 maximum square spot areas and complete all surgery.(0: unsatisfied; 5: very Satisfied)
Operating time | From beginning of the operation to the end of the operation with 10 maximum square spot areas;about ten seconds
  Operating time of 10 maximum square spot areas.

CONTACTS AND LOCATIONS:
Overall Officials: Lv Kaiyang, doctor, Principal Investigator — Changhai Hospital
Locations (1):
- HTC Vive, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gold MH, Berman B, Clementoni MT, Gauglitz GG, Nahai F, Murcia C. Updated international clinical recommendations on scar management: part 1--evaluating the evidence. Dermatol Surg. 2014 Aug;40(8):817-24. doi: 10.1111/dsu.0000000000000049. PMID 25068543
- [Result] Gold MH, McGuire M, Mustoe TA, Pusic A, Sachdev M, Waibel J, Murcia C; International Advisory Panel on Scar Management. Updated international clinical recommendations on scar management: part 2--algorithms for scar prevention and treatment. Dermatol Surg. 2014 Aug;40(8):825-31. doi: 10.1111/dsu.0000000000000050. PMID 25068544
- [Result] Manstein D, Herron GS, Sink RK, Tanner H, Anderson RR. Fractional photothermolysis: a new concept for cutaneous remodeling using microscopic patterns of thermal injury. Lasers Surg Med. 2004;34(5):426-38. doi: 10.1002/lsm.20048. PMID 15216537
- [Result] Anderson RR, Donelan MB, Hivnor C, Greeson E, Ross EV, Shumaker PR, Uebelhoer NS, Waibel JS. Laser treatment of traumatic scars with an emphasis on ablative fractional laser resurfacing: consensus report. JAMA Dermatol. 2014 Feb;150(2):187-93. doi: 10.1001/jamadermatol.2013.7761. PMID 24336931
- [Result] Hoffman HG, Chambers GT, Meyer WJ 3rd, Arceneaux LL, Russell WJ, Seibel EJ, Richards TL, Sharar SR, Patterson DR. Virtual reality as an adjunctive non-pharmacologic analgesic for acute burn pain during medical procedures. Ann Behav Med. 2011 Apr;41(2):183-91. doi: 10.1007/s12160-010-9248-7. PMID 21264690
- [Result] Wang HB, Fang Y, Yu WR. [Advancement in the research of fractional carbon dioxide laser in treating burn scars]. Zhonghua Shao Shang Za Zhi. 2012 Dec;28(6):465-7. Chinese. PMID 23327918
- [Result] Gallant J, Smith R, Wynn J, Vazquez E. 2012 HIV Drug Guide. Posit Aware. 2012 Mar-Apr;24(2):15-7, 22, 24-57 passim. No abstract available. PMID 22558746